CLINICAL TRIAL: NCT01293695
Title: Hypnosis For Hot Flashes Among Postmenopausal Women in a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Gary R. Elkins, PhD, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 194610; 5U01AT004634 (NIH)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-07

CONDITIONS: Hot Flashes
Keywords: hot flashes; post menopausal women; skin conductance monitors; hypnosis; hypnotizability
MeSH Terms: conditions — Hot Flashes | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypnosis (Active Comparator): Receives 5 weeks of hypnotic relaxation therapy
  Interventions: Behavioral: Hypnosis
- Structured Attention (Placebo Comparator): Meets with therapist for five weekly sessions, but receives no hypnotic relaxation therapy
  Interventions: Other: Structured attention

INTERVENTIONS:
Behavioral: Hypnosis — Hypnosis relaxation in five weekly sessions
  Other Names: Hypnotic relaxation therapy; Hypnosis relaxation; Hypnotic intervention; Hypnosis intervention
  Arms: Hypnosis
Other: Structured attention — Meets with therapist for five weekly sessions and receives structured attention/supportive counseling, but receives no hypnotic relaxation therapy
  Other Names: Placebo Comparator
  Arms: Structured Attention

SUMMARY:
This study is designed to determine the effect of a Hypnosis Intervention on reducing hot flash frequency (perceived impact vs. physiologically measured impact), severity and daily interference in post-menopausal women. It is felt that the Hypnosis Intervention will result in significantly lower hot flash frequency, severity and daily interference scores (perceived impact vs. physiologically measured impact) versus Structured-Attention Control.

DETAILED DESCRIPTION:
The aging population of the United States and findings from the Women's Health Initiative that indicate a shift in the risk/benefits balance of hormone therapy have created a growing interest in alternative treatments for hot flashes. Hot flashes are among the most severe and frequent symptoms experienced by women during menopause. Over 66% of post-menopausal women experience hot flashes. As a result, there is a pressing need for safe and effective treatments for hot flashes. Hypnosis is one mind-body therapy that seems particularly promising for treating hot flashes.

However, the treatment effectiveness of hypnosis in reducing physiologically measured (i.e. physiologically measured impact) hot flashes with post-menopausal women has yet to be established relative to a Structured-Attention Control. This is a critical step to further investigate the intervention and to determine if hypnosis reduces the symptoms (i.e. the number of physiological hot flashes) or only the women's perception of symptoms.

Also, the physiologic mechanism by which hypnosis may operate in reducing hot flashes is not known. The present study will compare hypnosis to a Structured-Attention Control in reducing hot flashes (perceived and physiologically monitored) in post-menopausal women in a randomized clinical trial.

Innovations of this study are that it will be the first full scale test of hypnosis for hot flashes; one of the first studies to examine both perceived impact and physiologically measured impact of a mind-body intervention for hot flashes using state-of-the-art 24 hour ambulatory physiological monitoring; the first study to examine the effect of hypnosis for hot flashes on cortisol; and the first investigation of the role of cognitive expectancies in treatment of hot flashes in comparison to a Structured-Attention Control.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal as defined by:

  1. no menstrual period in the past 12 months;
  2. no menstrual period in the past 6 months and a medically documented history of FSH level greater than 40; or
  3. women who have had a bilateral oophorectomy.
* A self-reported history of a minimum of 7 hot flashes per day or 50 hot flashes per week at baseline.
* Age over 18 years and ability to give her own consent for participation in the study.
* Have discontinued other putative therapies for hot flashes for at least one month prior to enrollment
* Ability to attend weekly sessions.

Exclusion Criteria:

* Receiving other simultaneous treatment for hot flashes.
* Using any CAM (Complementary and Alternative Medicine) treatments for vasomotor symptoms • Any medical or psychiatric condition that in the opinion of the investigator puts the participant at potential risk during the study.
* Currently using hypnosis for any reason.
* Inability to speak or understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2007-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R Elkins, Ph.D., Principal Investigator — Baylor University
Locations (1):
- Mind-Body Medicine Research Lab-Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts RL, Rhodes JR, Elkins GR. Effect of Hypnosis on Anxiety: Results from a Randomized Controlled Trial with Women in Postmenopause. J Clin Psychol Med Settings. 2021 Dec;28(4):868-881. doi: 10.1007/s10880-021-09810-3. Epub 2021 Aug 17. PMID 34403019
- [Derived] Elkins GR, Fisher WI, Johnson AK. Hypnosis for hot flashes among postmenopausal women study: a study protocol of an ongoing randomized clinical trial. BMC Complement Altern Med. 2011 Oct 11;11:92. doi: 10.1186/1472-6882-11-92. PMID 21989181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from December, 2008 to April, 2012. Participants were recruited by using fliers, mailings, billboard advertising and word-of-mouth. Local clinics were also visited and informative materials were left with physicians.
Groups:
- Structured Attention: Meets with therapist for five weekly sessions, but receives no hypnotic relaxation therapy
  Structured Attention: Meets for five weekly sessions for discussion on hot flashes; no hypnosis
Period: Overall Study
Arm/Group | Hypnosis | Structured Attention
Started | 93 | 94
Completed | 78 | 87
Not Completed | 15 | 7
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Lost to Follow-up | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Hypnosis: Receives 5 weeks of hypnotic relaxation therapy (HRT)
  Hypnosis: Hypnosis relaxation in five weekly sessions
- Total: Total of all reporting groups
Arm/Group | Hypnosis | Structured Attention | Total
Number analyzed (Participants) | 93 | 94 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 87 | 171
  >=65 years | 9 | 7 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 94 | 187
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 2 | 3 | 5
  Asian | 1 | 0 | 1
  African American | 20 | 11 | 31
  Hispanic | 6 | 6 | 12
  White | 64 | 74 | 138
Region of Enrollment [Number; unit: participants]
  United States | 93 | 94 | 187
Marital Status [Number; unit: participants]
  Married | 57 | 65 | 122
  Divorced | 8 | 10 | 18
  Separated | 5 | 5 | 10
  Single | 19 | 12 | 31
  Widowed | 4 | 2 | 6
Education [Number; unit: participants]
  Less than High School | 10 | 6 | 16
  High School Diploma | 26 | 26 | 52
  College, non degree | 20 | 20 | 40
  Associate Degree | 12 | 12 | 24
  Bachelor's Degree | 14 | 22 | 36
  Graduate Degree | 11 | 8 | 19
Hot Flash Frequency [Mean (Standard Deviation); unit: hot flashes per week] — Hot flash frequency and hot flash severity were obtained using the Hot Flash Symptoms Diary. Participants recorded their hot flashes over seven days marking each hot flash (frequency) and rating the severity of each as mild (1), moderate (2), severe (3), and very severe (4).
  hot flashes per week | 75.26 (2.82) | 75.21 (3.11) | 75.24 (2.97)
Hot Flash Score [Mean (Standard Deviation); unit: units on a scale] — Hot Flash Score is a product of frequency of hot flashes × severity of hot flashes, which could range from 0 (best possible outcome) to infinity (worst possible outcome).
  Hot flash frequency and hot flash severity were obtained using the Hot Flash Symptoms Diary. Participants recorded their daily hot flashes marking each hot flash (frequency) and rating the severity of each as mild (1), moderate (2), severe (3), and very severe (4).
  The values presented represent the average of daily hot flash scores.
  units on a scale | 24.43 (1.02) | 22.94 (1.23) | 23.69 (1.13)
Biolog Hot Flash Monitor (physiological measure) [Mean (Standard Deviation); unit: micro Siemens] — As a secondary outcome, hot flashes were measured using a Biolog ambulatory recorder. Skin conductance was expressed in micro Siemens (0 to infinity) and the final value was obtained by averaging the recorded skin conductance for a period of 24 hours. Lower skin conductance measure indicates less sweating.
  micro Siemens | 10.41 (1) | 8.85 (.75) | 9.63 (.88)
Hot Flash Related Daily Interference Scale (HFRDIS) [Mean (Standard Deviation); unit: units on a scale] — This questionnaire was used to measure the effects of hot flashes on women as they go about their daily activities. Answers on the scale can range 0 (Do Not Interfere) to 10 (Completely Interfere). The total score was computed by averaging the subjective ratings over the 10 items. A lower score indicates better outcome.
  units on a scale | 5.87 (.23) | 5.75 (.24) | 5.81 (24)
Pittsburg Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: units on a scale] — The Pittsburg Sleep Quality Index (PSQI) is a self-report inventory designed to measure sleep quality. The participants self rated their sleep quality over seven areas of sleep.The questions about sleep quality are answered on a 0-3 scale with higher scores indicating greater sleep pathology. The global score was determined by summing the raw scores of the seven sleep components. The global score can range from 0 - 21 and total scores above 5 are normally considered indicative of poor sleep quality.
  units on a scale | 11.69 (.56) | 11.89 (.48) | 11.79 (.52)

OUTCOME MEASURES:

1. Primary Outcome: Hot Flash Frequency
Description: The Hot Flash Symptoms Diary was used to measure hot flash frequency. Participants recorded their hot flashes over seven days by daily frequency and severity. This instrument provides a measure of hot flash frequency and hot flash score (product of frequency x severity).
Time Frame: 6 Weeks and 12 Weeks
Measure: Mean (Standard Deviation); unit: hot flashes per week
Groups:
- Hypnosis: Received 5 weeks of hypnotic relaxation therapy
  Hypnosis: Hypnosis relaxation in five weekly sessions. Weekly hot flash scores were averaged.
Arm/Group | Hypnosis | Structured Attention
Number analyzed (Participants) | 78 | 87
hot flashes per week
  Week 6 | 27.19 (2.48) | 68.26 (3.10)
  Week 12 | 19.44 (1.96) | 62.32 (3.43)

2. Primary Outcome: Hot Flash Score
Description: Hot Flash Score is a product of frequency of hot flashes × severity of hot flashes, which could range from 0 (best possible outcome) to infinity (worst possible outcome).
  Hot flash frequency and hot flash severity were obtained using the Hot Flash Symptoms Diary. Participants recorded their daily hot flashes marking each hot flash (frequency) and rating the severity of each as mild (1), moderate (2), severe (3), and very severe (4).
  The values presented represent the average of daily hot flash scores.
Time Frame: 6 Weeks and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hypnosis: Receives 5 weeks of hypnotic relaxation therapy
  Hypnosis: Hypnosis relaxation in five weekly sessions. Weekly hot flash scores were averaged.
Arm/Group | Hypnosis | Structured Attention
Number analyzed (Participants) | 78 | 87
units on a scale
  Week 6 | 6.71 (.79) | 21.03 (1.15)
  Week 12 | 4.61 (.56) | 19.41 (1.36)

3. Secondary Outcome: Sternal Skin Conductance Monitor Used to Physiologically Measure Skin Moisture
Description: As a secondary outcome, hot flashes were measured using a Biolog ambulatory recorder. Skin conductance was expressed in micro Siemens (0 to infinity) and the final value was obtained by averaging the recorded skin conductance for a period of 24 hours. Lower skin conductance measure indicates less sweating.
Time Frame: 6 Weeks and 12 Weeks
Population: Analysis was conducted on all available physiological data to determine hot flash frequency. Data was missing for 29 participants in the hypnosis group and 17 participants in the structured attention group.
Measure: Mean (Standard Deviation); unit: Micro Siemens
Arm/Group | Hypnosis | Structured Attention
Number analyzed (Participants) | 49 | 70
Micro Siemens
  Week 6 | 6.15 (.81) | 9.48 (.87)
  Week 12 | 4.49 (.59) | 7.97 (.70)

4. Secondary Outcome: Pittsburg Sleep Quality Index (PSQI)
Description: The Pittsburg Sleep Quality Index (PSQI) is a self-report inventory designed to measure sleep quality. The participants self rate their sleep quality over seven areas of sleep.The questions about sleep quality are answered on a 0-3 scale with higher scores indicating greater sleep pathology. The global score is determined by summing the raw scores of the seven sleep components. The global score can range from 0 - 21 and total scores above 5 are normally considered indicative of poor sleep quality.
Time Frame: 6 Weeks and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypnosis | Structured Attention
Number analyzed (Participants) | 78 | 87
units on a scale
  Week 6 | 6.10 (.47) | 10.85 (.51)
  Week 12 | 5.42 (.47) | 10.66 (.55)

5. Primary Outcome: Hot Flash Related Daily Interference Scale (HFRDIS)
Description: This questionnaire is used to measure the effects of hot flashes on women as they go about their daily activities. Answers on the scale can range 0 (Do Not Interfere) to 10 (Completely Interfere). The total score was computed by averaging the subjective ratings over the 10 items. A lower score indicates better outcome.
Time Frame: 6 Weeks and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypnosis | Structured Attention
Number analyzed (Participants) | 78 | 87
units on a scale
  Week 6 | 1.85 (.21) | 4.71 (.27)
  Week 12 | 1.05 (.20) | 4.43 (.28)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 12 weeks. (i.e.: weekly from baseline to 12 week follow-up)
Description: Adverse events were assessed at each session by participant self-report.
Arm/Group | Hypnosis | Structured Attention
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/94
Other Adverse Events (participants affected / at risk) | 13/93 | 12/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hypnosis (N=93) | Structured Attention (N=94)
Skin irritation (Skin and subcutaneous tissue disorders) | 13 | 12 — mild skin irritation from the skin conductance monitor electrode adhesive, requiring no medical intervention to resolve.

LIMITATIONS AND CAVEATS:
limitations: results may not generalize to all women with hot flashes

* some hot flashes occur at other times than during the climacteric
* self-selection bias (predispositions to mind-body therapy)
* population was largely caucasian

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No